CLINICAL TRIAL: NCT06685757
Title: A Double-Blind, Placebo-Controlled, Multicenter, Randomized Phase 3 Trial Evaluating the Efficacy and Safety of Felzartamab in Kidney Transplant Recipients With Late Antibody-Mediated Rejection (AMR)
Brief Title: A Study to Learn More About the Effects and Safety of Felzartamab Infusions in Adults With Kidney Transplants Who Have Antibody-Mediated Rejection (AMR)
Acronym: TRANSCEND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 299AR301; 2024-519095-66-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Antibody-mediated Rejection
Keywords: AMR; Felzartamab; Kidney Transplant
MeSH Terms: interventions — felzartamab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a 2-part trial; Part A will be randomized and placebo-controlled, and Part B will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Felzartamab (Experimental)
  Interventions: Drug: Felzartamab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Felzartamab — Participants will receive felzartamab by intravenous infusion.
  Other Names: MOR202; MOR03087; TJ202; HIB202; BIIB148
  Arms: Felzartamab
Drug: Placebo — Participants will receive 0.9% saline solution by intravenous infusion.
  Arms: Placebo

SUMMARY:
In this study, researchers will learn more about the use of felzartamab in kidney transplant patients who have antibody-mediated rejection, also known as AMR. Kidney transplants can save lives for people with kidney failure. But even after a successful transplant, the body's immune system can sometimes attack the new kidney.

Antibody-mediated rejection (AMR) is when a person's immune system attacks a transplanted organ, like a new kidney. In the person receiving the transplant, their immune system creates specific antibodies. Antibodies are proteins that help the body fight infections. In people with AMR, these antibodies mistakenly see the new organ as a threat and damage its blood vessels. This can cause the new organ to fail.

In this study, researchers will learn more about how a study drug called felzartamab affects people with AMR. Felzartamab is a monoclonal antibody, which means it is an antibody made in a laboratory. Felzartamab can target immune cells that produce antibodies, helping to lower their buildup in the kidneys. The main goal of this study is to compare how felzartamab works in participants with kidney transplants who experience AMR compared to a placebo. A placebo is something that looks like the study drug but does not contain any medicine. A placebo is also given in the same way as the study drug. All participants in this study will have active AMR or AMR that has lasted for at least 6 months after their kidney transplant.

The main question that researchers want to answer is:

• How many participants have biopsy results showing that their transplanted kidney tissue looks normal or near normal after 24 weeks of treatment?

Researchers will also learn about:

* How long it takes before the participants' disease gets worse
* How long the participants' urine protein levels stay low
* Kidney biopsy scores to check for blood vessel inflammation at 6 months and 1 year
* How many people have no blood vessel inflammation at these times
* Changes in donor deoxyribonucleic acid (DNA) levels in blood from the start of treatment
* Biopsy test scores for signs of rejection and inflammation at 6 months and 1 year
* Changes in kidney function from the start of treatment
* How many people have biopsy results showing their kidney tissue looks normal again
* How long the transplanted kidney keeps working
* How many participants have medical problems during the study
* How many participants show signs of another type of kidney transplant rejection called T-cell-mediated rejection (TCMR) at Week 24 and Week 52
* How do results from vital signs, electrocardiograms (ECGs), and blood and urine tests change over time
* How felzartamab is processed by the body
* How many participants develop antibodies against felzartamab in the blood

The study will be done as follows:

* Participants will be screened to check if they can join the study. This will take up to 42 days.
* There will be 2 parts in this study.
* Part A of the study is "double blind." This means that neither the participants, study doctor, or site staff know if the participants received the study drug or a placebo. During Part A, participants will be randomized to receive up to 9 doses of either felzartamab or placebo.
* Part B of the study is "open label." This means that the participants, study doctor, and site staff know which study drug the participant is receiving. During Part B, all participants from Part A will receive up to 9 doses of felzartamab.
* All doses will be given through an "intravenous" infusion. This means it will be given into a vein. The dose the participants receive will depend on their body weight.
* Part A will last up to 24 weeks. Part B will last up to 28 weeks. In total, participants will have up to 21 study visits and will be in the study for about 1 year.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of felzartamab compared to placebo in kidney transplant recipients diagnosed with active or chronic active AMR.

The secondary objectives of this study are: Part A: To evaluate the efficacy of felzartamab compared to placebo through additional clinical endpoints; Part B: To summarize felzartamab efficacy at Week 52 in kidney transplant recipients diagnosed with active or chronic active AMR; Parts A and B: To evaluate the safety of felzartamab in kidney transplant recipients diagnosed with active or chronic AMR and to assess the pharmacokinetic (PK) profile and immunogenicity of felzartamab.

ELIGIBILITY:
Key Inclusion Criteria:

* Active or chronic active AMR (biopsy-confirmed) without TCMR per central reading, as defined by the Banff 2022 criteria.
* Kidney transplant at least 6 months prior to Screening visit (recipients of either living or deceased donors).
* Donor-specific antibody (DSA): Human leukocyte antigen (HLA) Class I and/or II antigen-specific DSA-positive (preformed and/or de novo DSA) as determined by the local laboratory's definition of positivity using singleantigen bead-based assays within 3 months prior to randomization.

Key Exclusion Criteria:

* Transplant: Blood type (ABO)-incompatible transplant.
* History of multiple organ transplants including en bloc and dual kidney transplants.
* Acute, rapid decline in renal function, defined as a participant likely to require renal replacement therapy within the subsequent 30 days as determined by the Investigator.
* Treatment: Prior AMR/TCMR treatment (with the exception of corticosteroids) within 3 months prior to randomization is excluded as listed below. Participants who received any of these treatments between 3 and 6 months prior to randomization must have both a renal biopsy (IC3) and DSA testing at least 6 weeks after completing (or stopping) treatment in order to confirm continuing AMR and to determine eligibility:

  1. Intravenous or subcutaneous immunoglobulin (IVIg or subcutaneous immunoglobulin [SCIg]) or PLEX.
  2. Complement system inhibitors (e.g., eculizumab).
  3. Proteasome inhibitors (e.g., bortezomib).
  4. Tocilizumab.
  5. Any B cell-depleting therapy (including anti-Cluster of Differentiation 20 [CD20] agents [e.g., rituximab]) within 3 months prior to randomization.
  6. Any other investigational agent within 3 months or 5 half-lives (whichever is longer) of randomization.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants Who Achieve Biopsy-proven Histologic Resolution (BPHR) | Week 24

SECONDARY OUTCOMES:
Part A: Microvascular Inflammation (MVI) Score | Week 24
Part A: Percentage of Participants Who Achieve an MVI Score of 0 | Week 24
Part A: Change from Baseline in Donor-derived Cell-free DNA (dd-cfDNA) | Baseline, Week 24
Part A: Biopsy-based Transcript Composite Score for AMR/MVI | At Week 24
Part A: Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 24
Part B: Percentage of Participants Who Achieve BPHR | Weeks 24 and 52
Part B: MVI Score | Weeks 24 and 52
Part B: Percentage of Participants Who Achieve an MVI Score of 0 | Weeks 24 and 52
Part B: Change from Baseline in dd-cfDNA | Baseline, Weeks 24 and 52
Part B: Biopsy-based Transcript Composite Score for AMR/MVI | At Week 52
Part B: Change from Baseline in eGFR | Baseline, Weeks 24 and 52
Part B: Time to All-cause Allograft Loss | Up to Week 52
Parts A and B: Number of Participants with Adverse Events | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Number of Participants with Clinically Significant Laboratory Abnormalities | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Number of Participants with Clinically Significant Vital Signs Abnormalities | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Number of Participants with Clinically Significant ECG Abnormalities | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Percentage of Participants with T Cell-mediated Rejection (TCMR) by Biopsy | Weeks 24 and 52
Parts A and B: Felzartamab Serum Concentration | Up to Week 52
Parts A and B: Number of Participants with Anti-drug Antibodies (ADAs) against Felzartamab | Baseline, up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (57):
- United States (27):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Providence Healthcare, Orange, California
  - Loma Linda, San Bernardino, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Cooperman Barnabas Medical Center, West Orange, New Jersey
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Penn Medicine - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Instituto de Trasplante y Alta Complejidad (ITAC), Cdad, Autónoma de Buenos Aires, Argentina
- Australia (4):
  - Royal Melbourne Hospital, Parkville VIC, Australia
  - Westmead Hospital, Sydney, New South Wales
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Princess Alexandra Hospital, Woolloongabba
- Medical University of Vienna, Spitalgasse, Vienna, Austria
- Brazil (4):
  - Santa Casa de Misericordia de Porto Alegre - Hospital Dom Vicente Scherer, Centro Histórico, Porto Alegre - RS
  - Hospital de Base da Faculdade de Medicina de São José do Rio Preto, Vila São José, São José Do Rio Preto
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, Cerqueira César, São Paulo
  - Fundação Oswaldo Ramos - Hospital do Rim (HRIM), Vila Clementino, São Paulo
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - The University of British Columbia (UBC)/St. Paul's Hospital part of Providence Health Care, Vancouver, British Columbia
  - McGill University, Montreal, Quebec
- France (4):
  - CHU Lyon Hôpital Edouard Herriot, Bordeaux
  - CHU Grenoble Alpes Hôpital Michallon, La Tronche
  - Hospices Civils de Lyon - Hôpital Édouard Herriot, Lyon
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hôpital de Rangueil, Toulouse
- Germany (4):
  - Charite University, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Regensburg, Regensburg
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Spain (5):
  - Hospital Clinic de Barcelona, Calle Villarroel, Barcelona
  - Hospital del Mar, Ciutat Vella, Barcelona
  - Hospital Universitario Vall d'Hebron, Horta-Guinardó, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (2):
  - University Hospital Basel, Petersgraben, Basel
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Bohmig GA, Akifova A, Budde K. World Transplant Congress 2025 Highlights: Immunosuppression. Transplantation. 2026 Feb 1;110(2):e356-e362. doi: 10.1097/TP.0000000000005569. Epub 2025 Dec 23. PMID 41430762